CLINICAL TRIAL: NCT05054946
Title: The Effect of Laparoscopic Surgery on Ovarian Reserve According to Cyst Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Principal Investigator, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/056
Record Dates: First submitted 2021-09-19; First posted 2021-09-23 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cysts
Keywords: ovarian reserve; anti-mullerian hormone; ovarian cyst
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endometrioma (Active Comparator): Participants who will have endometrioma after histopathological evaluation.
  Interventions: Procedure: Laparoscopic cystectomy
- Mature cystic teratoma (dermoid cyst) (Active Comparator): Participants who will have mature cystic teratoma (dermoid cyst) after histopathological evaluation.
  Interventions: Procedure: Laparoscopic cystectomy
- Serous or mucinous cystadenoma (Active Comparator): Participants who will have serous or mucinous cystadenoma after histopathological evaluation.
  Interventions: Procedure: Laparoscopic cystectomy

INTERVENTIONS:
Procedure: Laparoscopic cystectomy — All surgeries will be performed under general anesthesia by laparoscopically.

SUMMARY:
The aim of our study is to compare the effect of laparoscopic ovarian cystectomy on ovarian reserve in terms of different cyst types.

DETAILED DESCRIPTION:
Participants who will be treated surgically for ovarian cysts will be included in the study. Anti-Mullerian Hormone (AMH) levels of the participants will be investigated before the surgery and 6 months after the surgery. All surgeries will be performed under general anesthesia laparoscopically. After histopathological evaluation, the participants will be divided into three groups; Group 1: Endometrioma, Group 2: Mature cystic teratoma (Dermoid cyst) and Group 3: Serous or mucinous cystadenoma.

A total of fifty-five women will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* no ovarian surgery before

Exclusion Criteria:

* Endocrinological pathologies
* Suspicion of malignancy in preoperative laboratory and ultrasonographic evaluations
* Detection of malignancy in histopathological examination

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in AMH Level | 6 months
  AMH levels of the participants will be investigated before the surgery and 6 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sabahattin Anil Ari, MD, Principal Investigator — Ege University
Locations (1):
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No